CLINICAL TRIAL: NCT03736083
Title: Introducing Continuous Glucose Monitoring Technology at Diagnosis in Pediatric Type 1 Diabetes: A Proof of Concept Study
Brief Title: Introducing CGM at Type 1 Diabetes Diagnosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA approval not obtained.
Sponsor: University of Florida (Other)
Collaborators: Diabetes Action Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201802031 -A; OCR19017 (Other: UF ID)
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Type1diabetes; Hypoglycemia
Keywords: glucose monitoring; glycemic control
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Intervention Model Description: The study team will enroll 52 consecutive new onset type 1 diabetes patients and stratify the subjects into two groups, age 4-10 vs 11-17, aiming for 26 subjects in each group. Participants will be randomized to one of the two groups using blocked randomization with random block sizes of 2 and 4, stratified by age (4-10 vs. 11-17).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Freestyle Libre Group (Active Comparator): Freestyle Libre Group: Participants will use the Freestyle Libre flash glucose monitoring system throughout the study for 2-3 months.
  Interventions: Device: Freestyle Libre Blood Glucose Monitor
- Control Group (standard diabetes care) (No Intervention): This group will receive standard care. At the around 1 week and 2 month visits, control group subjects will use a blinded Freestyle Libre Pro to provide data that can be used to compare glucose variability between groups. The Libre sensor will allow the study team to measure glucose values but the subjects will not have access to this information for management/treatment decisions and usual diabetes care will be unaffected. The Freestyle Libre Pro last 14 days, can be activated in clinic, and the sensor can be returned in person or via mail where the investigators will download the data.

INTERVENTIONS:
Device: Freestyle Libre Blood Glucose Monitor — The intervention arm of this study will begin using the Freestyle Libre glucose monitor within 2 weeks of their diabetes diagnosis
  Arms: Freestyle Libre Group

SUMMARY:
Diabetes technology is changing and has quickly become an integral part of diabetes care and management. The study team plans to study the effects of introducing technology to newly diagnosed type 1 diabetes patients. The investigators hypothesize that early access to continuous glucose monitoring (CGM) technology will potentially improve satisfaction scores, hemoglobin A1c, glycemic control, reduce hypoglycemia, and ease the burden of disease when compared to new onset patients who receive standard of care access to CGM.

DETAILED DESCRIPTION:
Abstract: Diabetes technology is changing and has quickly become an integral part of diabetes care and management. Typically, patients will need to wait months due to paperwork, insurance, and logistical issues before utilizing these technologies. With this project, the investigators plan to study the effects of introducing technology to newly diagnosed type 1 diabetes patients. It is hypothesized that early access to flash continuous glucose monitoring (CGM) technology will improve scores in diabetes's measures. The primary outcome with be the parent version of the Diabetes Treatment Satisfaction Questionnaire (DTSQ). Secondary outcomes will include other diabetes measures such as DTSQ teen version, Hypoglycemia Fear Survey (HFS)- Parent and child version, Diabetes Distress Survey (DDS)-parent version, PedsQL- parent and child versions. The study team will also look at other diabetes outcomes including A1c, time in range, and reduction in hypoglycemia.

Background: Type 1 diabetes is a complex disease requiring newly diagnosed pediatric patients and families to learn how to check blood glucoses, inject insulin, count carbohydrates, treat hypoglycemia/hyperglycemia, and perform many other complex tasks, all within the first few days after diagnosis.

Continuous glucose monitors (CGMs) and flash glucose monitors have emerged as important diabetes technologies towards providing improved care and easing the burden of disease. These technologies are most typically introduced to families in the outpatient setting 2-3 months following diagnosis due to logistical issues related to insurance coverage.

Barriers to access include requirements for insurance prior authorization, lack of immediate availability at local pharmacies, need for patient training, and the historical bias towards requiring finger stick glucose monitoring as the basis for diabetes management. Despite these barriers, the data supports the observation that CGM technology provides for better understanding of diabetes, improved quality of life for parents and children, reduced frequency of hypoglycemia, and improved A1c.

This project will potentially show the feasibility of introducing these technologies at diagnosis. New onset type 1 diabetes patients will be randomized to receive either a Freestyle Libre flash glucose monitoring system immediately at diagnosis or to delayed use of CGM (standard of care).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus

Exclusion Criteria:

* No diagnosis of type 1 diabetes mellitus

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Change in Diabetes Treatment Satisfaction Questionnaire- Parent version | 2 weeks,3 months, and 12 months
  Survey for Diabetes treatment satisfaction: 14 question survey with each question scaled from 0-6; with 0 being 'very dissatisfied' and 4 being 'very satisfied'

SECONDARY OUTCOMES:
Change in Diabetes Treatment Satisfaction Questionnaire- Teen version | 2 weeks,3 months, and 12 months
  Survey for Diabetes treatment satisfaction: 12 question survey with each question scaled from 0-6; with 0 being 'very dissatisfied' and 6 being 'very satisfied
Change in Pediatric Quality of Life Survey- Parent and child versions | 2 weeks,3 months, and 12 months
  Survey for Pediatric quality of life: 33 question survey with each question scaled from 0-4; with 0 being 'never to 4 being 'almost always'
Change in Problem Areas in Diabetes survey | 2 weeks,3 months, and 12 months
  Survey for diabetes specific distress: mean item score or 0 - 1.9 should be considered "little or no distress," a mean item score between 2.0 - 2.9 should be considered 'moderate distress,' and a mean item score > 3.0 should be considered 'high distress.'
Change in Hypoglycemia Fear Survey - Parent and Child Versions | 2 weeks,3 months, and 12 months
  Survey for fear associated with hypoglycemia: 26 question survey with each question scaled from 0-4; with 0 being 'never' and 4 being 'almost always'
Change in Diabetes Distress Survey- Parent version | 2 weeks,3 months, and 12 months
  The PARENT DDS yields a total diabetes distress score plus 4 subscale scores, each addressing a different kind of distress. To score, simply sum the patient's responses to the appropriate items and divide by the number of items in that scale.
  Current research suggests that a mean item score or 0 - 1.9 should be considered "little or no distress," a mean item score between 2.0 - 2.9 should be considered 'moderate distress,' and a mean item score > 3.0 should be considered 'high distress.'
Change in Glycemic control measured by A1c | 3 and 12 months
  Measurement of A1c

OTHER OUTCOMES:
Number of flash glucose measurements at the intervention arm | 3 months
  # of flash measurements provided by the freestyle reader
Number of glucose measurements of the control arm | 3 months
  # of glucose readers based on there glucose meter download
Percentage of glucose sensor readings within the range of 70 to 180 mg/dl | 3 months
  Data by Freestyle libre readings
Percentage of glucose sensor readings below 80 mg/dl | 3 months
  Data by Freestyle libre readings
Percentage of glucose sensor readings above 180 mg/dl | 3 months
  Data by Freestyle libre readings

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hiers, MD, Principal Investigator — University of Florida

REFERENCES:
- [Background] Bolinder J, Antuna R, Geelhoed-Duijvestijn P, Kroger J, Weitgasser R. Novel glucose-sensing technology and hypoglycaemia in type 1 diabetes: a multicentre, non-masked, randomised controlled trial. Lancet. 2016 Nov 5;388(10057):2254-2263. doi: 10.1016/S0140-6736(16)31535-5. Epub 2016 Sep 12. PMID 27634581
- [Background] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group. Effectiveness of continuous glucose monitoring in a clinical care environment: evidence from the Juvenile Diabetes Research Foundation continuous glucose monitoring (JDRF-CGM) trial. Diabetes Care. 2010 Jan;33(1):17-22. doi: 10.2337/dc09-1502. Epub 2009 Oct 16. PMID 19837791
- [Background] Shapiro JB, Vesco AT, Weil LEG, Evans MA, Hood KK, Weissberg-Benchell J. Psychometric Properties of the Problem Areas in Diabetes: Teen and Parent of Teen Versions. J Pediatr Psychol. 2018 Jun 1;43(5):561-571. doi: 10.1093/jpepsy/jsx146. PMID 29267939
- [Background] Barnard K, Thomas S, Royle P, Noyes K, Waugh N. Fear of hypoglycaemia in parents of young children with type 1 diabetes: a systematic review. BMC Pediatr. 2010 Jul 15;10:50. doi: 10.1186/1471-2431-10-50. PMID 20633252
- [Background] Gonder-Frederick L, Nyer M, Shepard JA, Vajda K, Clarke W. Assessing fear of hypoglycemia in children with Type 1 diabetes and their parents. Diabetes Manag (Lond). 2011;1(6):627-639. doi: 10.2217/DMT.11.60. PMID 22180760
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Background] Varni JW, Burwinkle TM, Jacobs JR, Gottschalk M, Kaufman F, Jones KL. The PedsQL in type 1 and type 2 diabetes: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales and type 1 Diabetes Module. Diabetes Care. 2003 Mar;26(3):631-7. doi: 10.2337/diacare.26.3.631. PMID 12610013
- [Background] Markowitz JT, Volkening LK, Butler DA, Laffel LM. Youth-Perceived Burden of Type 1 Diabetes: Problem Areas in Diabetes Survey-Pediatric Version (PAID-Peds). J Diabetes Sci Technol. 2015 Apr 24;9(5):1080-5. doi: 10.1177/1932296815583506. PMID 25910541